CLINICAL TRIAL: NCT07112963
Title: "Comparison of the Effects of Resin Infiltrant, Fluoride Varnish, and the Combined Application of Resin Infiltrant and Fluoride Varnish on Primary Molars in the Treatment of Proximal Non-Cavitated Carious Lesions in Children."
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sacide Duman (Other)
Responsible Party: Sponsor-Investigator, Sacide Duman, Associate Professor, Inonu University
Organization: Inonu University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022/80
Record Dates: First submitted 2025-08-01; First posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Dental Caries; Tooth Demineralization; Pediatric Dentistry; Molar, Deciduous
Keywords: Fluoride varnish; Proximal caries; Pediatric dentistry; Resins, Synthetic
MeSH Terms: conditions — Dental Caries; Tooth Demineralization

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned into three parallel groups: fluoride varnish only, resin infiltration only, and a combination of resin infiltration and fluoride varnish. Each group received its designated intervention, and no crossover occurred between groups.
Masking Description: This study was conducted as an open-label trial. Neither participants, investigators, nor outcome assessors were blinded to group assignments due to the nature of the interventions.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Fluoride Varnish Group (Active Comparator): Participants in this group receive only fluoride varnish applications according to standard clinical protocols. The treatment aims to remineralize early proximal carious lesions and prevent progression.
  Interventions: Drug: Fluoride Varnish
- Resin Infiltration Group (Experimental): Participants in this group receive resin infiltration treatment alone, applied following manufacturer guidelines and standardized procedures, aiming to arrest or reverse early enamel carious lesions.
  Interventions: Drug: Fluoride Varnish
- Resin Infiltration + Fluoride Varnish Group (Experimental): Participants in this group receive a combined intervention of resin infiltration followed by fluoride varnish application. The combined treatment is intended to maximize caries arrest and promote remineralization of proximal lesions.
  Interventions: Drug: Fluoride Varnish

INTERVENTIONS:
Drug: Fluoride Varnish — Application of fluoride varnish to proximal surfaces of primary molars following standard clinical protocols to promote remineralization and arrest early carious lesions.
  Application of resin infiltrant material to proximal non-cavitated carious lesions in primary molars, performed according to manufacturer instructions to arrest lesion progression.
  Sequential application of resin infiltration followed by fluoride varnish on proximal surfaces of primary molars to maximize caries arrest and remineralization effects.
  Other Names: Resin Infiltration; Resin Infiltration and Fluoride Varnish Combination

SUMMARY:
Purpose:

This randomized controlled clinical trial aimed to compare the effectiveness of fluoride varnish, resin infiltrant, and their combination in treating superficial proximal carious lesions in primary molars of children aged 4 to 9 years.

Materials and Methods:

Twenty-six children with initial proximal caries (E1, E2, D1) on primary molars were randomly assigned to three groups: fluoride varnish only (F), resin infiltration only (RI), and resin infiltration combined with fluoride varnish (RI+F). Treatments were applied according to standardized protocols, and clinical and radiographic evaluations were conducted at 3, 6, 9, and 12 months.

DETAILED DESCRIPTION:
This randomized controlled clinical trial investigates the comparative effectiveness of fluoride varnish, resin infiltrant, and their combined use in managing superficial proximal carious lesions in primary molars of children aged 4 to 9 years. A total of 26 pediatric patients presenting with initial proximal caries lesions classified as E1, E2, and D1 levels were enrolled. Participants were randomly allocated into three groups: fluoride varnish only (F), resin infiltration only (RI), and a combination of resin infiltration with fluoride varnish (RI+F).

Interventions were applied according to standardized clinical protocols. Follow-up assessments, including clinical examinations and radiographic evaluations, were conducted at 3, 6, 9, and 12 months post-treatment to monitor lesion progression or regression. The primary outcome measure was the change in caries lesion status over time, evaluated through clinical and radiographic criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age between 4 and 9 years

Presence of initial proximal carious lesions (E1, E2, D1) on primary molars

Generally healthy children without systemic diseases

Consent obtained from parents or legal guardians

Exclusion Criteria:

* Cavitated or advanced proximal carious lesions

Known allergy to fluoride varnish or resin infiltrant materials

Systemic diseases affecting oral health or participation

Prior restorative treatment on the target teeth

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2023-10-04 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Caries Lesion Progression | 12 months
  The primary outcome is the clinical and radiographic assessment of proximal carious lesion progression or arrest in primary molars over a 12-month follow-up period. Lesion status will be evaluated at 3, 6, 9, and 12 months to determine treatment efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Inonu University, Faculty of Dentistry, Malatya, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
The individual participant data (IPD) from this study will be shared in a de-identified form. Data will be made available upon reasonable request to the corresponding author after publication of the primary results. Access will be granted following approval of a data use agreement and ethics compliance.

REFERENCES:
- [Background] Paris S, Meyer-Lueckel H. Infiltrants inhibit progression of natural caries lesions in vitro. J Dent Res. 2010 Nov;89(11):1276-80. doi: 10.1177/0022034510376040. Epub 2010 Aug 25. PMID 20739697
- [Background] Martignon S, Ekstrand KR, Gomez J, Lara JS, Cortes A. Infiltrating/sealing proximal caries lesions: a 3-year randomized clinical trial. J Dent Res. 2012 Mar;91(3):288-92. doi: 10.1177/0022034511435328. Epub 2012 Jan 17. PMID 22257664